CLINICAL TRIAL: NCT03457259
Title: The Clinical Efficacy of Midline Catheters for Intravenous Therapy: a Randomized, Controlled Study
Brief Title: The Clinical Efficacy of Midline Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Emma Bundgaard Nielsen, Medical student, Research student, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: midlineivauh18
Record Dates: First submitted 2018-02-13; First posted 2018-03-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Intravenous Catheters
Keywords: Midline catheter, peripheral venous catheter, central venous catheter, complication rate

STUDY DESIGN:
Intervention Model Description: 60 patients in each group, with a total of 2 groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midline (Active Comparator): Pt. will receive midline catheters. The outcomes will be registered and some patients will be examined once weekly for thrombosis with ultrasound.
  Interventions: Device: Midline
- Conventional (Active Comparator): Pt. will receive the conventional treatment (PVC and/or PICCline/CVC). The outcomes will be registered.
  Interventions: Device: PVC and/or PICCline

INTERVENTIONS:
Device: PVC and/or PICCline — Pt. will receive PVC and/or PICCline
  Other Names: Conventional catheterization
  Arms: Conventional
Device: Midline — Pt. will receive midline
  Other Names: Powerglide
  Arms: Midline

SUMMARY:
The study will evaluate the clinical efficacy of midline catheters compared to conventional treatment in patients with an expected intravenous therapy duration of more than 5 days. Patients will be randomized in a 1:1 ratio. The study will include 120 patient. Endpoints include insertion of CVSs, peripheral venous catheters, catheter patency and a number of possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Department of Infectious Disease or Department of Heart Disease.
* ≥18 years of age
* Expected requirement for iv. therapy >5 days from the day of enrolment as evaluated by a specialist in infectious diseases.
* Mentally competency

Exclusion Criteria:

* Lack of patient consent
* Requirement for a CVC before study eligibility screening or anticipation of an absolute indication for CVC inserted within 24 hours of screening
* Personnel for insertion of midline catheter not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Reducing the use of CVC and PVC | through study completion, an average of 7 month
  The fraction of patients requiring either a CVC - including PICC line - or require ≥ 4PVC insertions during the current admittance to the hospital, including follow-up intravenous therapy.

SECONDARY OUTCOMES:
Bloodsamples from catheter | through study completion, an average of 7 month
  Registration of number of blood samples taken from the midline catheter
Problems with catheter bloodsampling | through study completion, an average of 7 month
  Registration of aspiration problems during bloodsampling in midline catheters
Bloodsamples (conventional) | through study completion, an average of 7 month
  Registration of number of blood samples taken from conventional blood samples in both groups
Patient satisfaction | through study completion, an average of 7 month
  Patient satisfaction on NRS score, 0 is very unsatisfied and 10 is very satisfied
Nurse satisfaction | through study completion, an average of 7 month
  Nurse satisfaction on NRS score, 0 is very unsatisfied and 10 is very satisfied
Painscore | through study completion, an average of 7 month
  Accumulated NRS pain score for all IV catheter insertions. 0 is no pain and 10 is worst imaginable pain
Rescue catherizations 1 | through study completion, an average of 7 month
  Rescue PVC's inserted (midline group) (no)
Rescue catherizations 2 | through study completion, an average of 7 month
  Rescue central venous catheters including PICC line catheters inserted (no)
Time consumption | through study completion, an average of 7 month
  Total time of cauterization, (measured from the entrance in patient room, to the exit)
Catheter dwelltime | through study completion, an average of 7 month
  Time of catheter duration (hours)
Fluid | through study completion, an average of 7 month
  Accumulated fluids infused (L)
Treatment type | through study completion, an average of 7 month
  Type of medicine infused (all types)
Treatment amount | through study completion, an average of 7 month
  Amount of medicine infused (L)
Catheter related infections | through study completion, an average of 7 month
  Catheters removed due to suspected catheter-related infection (no)
Thrombosis 1 | through study completion, an average of 7 month
  Thrombi visible at the catheter tip (no)
Thrombosis 2 | through study completion, an average of 7 month
  Deep venous thrombosis of the ipsilateral arm (no)
Thrombosis 3 | through study completion, an average of 7 month
  Superficial venous thrombosis of the ipsilateral arm (midline group) (no)
Thrombosis 4 | through study completion, an average of 7 month
  Patients starting anti-thrombotic medicine due to thrombi generated by an IV catheter (no)
Catheter discontinuation | through study completion, an average of 7 month
  Reasons for replacing catheters (all types)
Insertion complication | through study completion, an average of 7 month
  Arterial punctures during catheter insertions (no)
Insertion complication 2 | through study completion, an average of 7 month
  haematomas during catheter insertions (no)
Insertion complication 3 | through study completion, an average of 7 month
  Misplaced catheters (no)
Neuropraxia | through study completion, an average of 7 month
  Post-procedure median nerve palsy/neuropraxia (midline group) (no)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Bundgaard, MS, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Anaesthesiology and Intensive Care East Section, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736